CLINICAL TRIAL: NCT01871571
Title: Phase II Trial Of Neoadjuvant Bevacizumab With Modified FOLFOX7 In Patients With Stage II And III Rectal Cancer
Brief Title: Bevacizumab, Fluorouracil, Leucovorin Calcium, and Oxaliplatin Before Surgery in Treating Patients With Stage II-III Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3R-12-2; NCI-2013-01069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ML28263; P30CA014089 (NIH)
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Mucinous Adenocarcinoma of the Rectum; Signet Ring Adenocarcinoma of the Rectum; Stage IIA Rectal Cancer; Stage IIB Rectal Cancer; Stage IIC Rectal Cancer; Stage IIIA Rectal Cancer; Stage IIIB Rectal Cancer; Stage IIIC Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (bevacizumab, mFOLFOX7) (Experimental): Patients receive bevacizumab IV over 30-90 minutes, oxaliplatin IV over 2 hours, leucovorin calcium IV, and fluorouracil IV continuously over 46-48 hours on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity. Within 6-8 weeks after treatment, patients undergo surgery.
  Interventions: Biological: bevacizumab; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well bevacizumab, fluorouracil, leucovorin calcium, and oxaliplatin before surgery works in treating patients with stage II-III rectal cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as fluorouracil, leucovorin calcium, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with fluorouracil, leucovorin calcium, and oxaliplatin may be an effective treatment for rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if six cycles of modified fluorouracil, leucovorin calcium, and oxaliplatin (mFOLFOX7) plus bevacizumab (Avastin) will yield complete pathologic response (cPR) of 25% or more in the primary tumor of patients with stage II and III rectal cancer.

SECONDARY OBJECTIVES:

I. To assess the rate of tumor regression (pathologic stage lower than clinical stage) after 6 cycles of mFOLFOX7 and bevacizumab in the primary rectal cancer.

II. To assess local recurrence rate over 3 years after 6 cycles of mFOLFOX7 and bevacizumab.

TERTIARY OBJECTIVES:

I. Correlation of the following marker with response (defined as CPR or down staging):

* Intratumoral Gene expression and germline polymorphism of genes involved in the vascular endothelial growth factor (VEGF) and VEGF independent pathways (VEGF, vascular endothelial growth factor receptor 1 [VEGFR1], VEGFR2, interleukin-8 [IL8], chemokine (C-X-C motif) receptor 2 [CXCR2], intercellular adhesion molecule [ICAM], VEGFR1 and VEGFR2, neuropilin 1 or 2 [NRP1,2], cluster of differentiation [CD] 44, aldehyde dehydrogenase [ALDH], leucine-rich repeats and immunoglobulin-like [LRIG].
* Circulating tumor cells (CTC) and VEGF-factor A (A) on the CTC.

II. Prediction of surgical resection margin by pretreatment magnetic resonance imaging (MRI).

OUTLINE:

Patients receive bevacizumab intravenously (IV) over 30-90 minutes, oxaliplatin IV over 2 hours, leucovorin calcium IV, and fluorouracil IV continuously over 46-48 hours on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity. Within 6-8 weeks after treatment, patients undergo surgery.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum in patients with no prior therapy who are candidate for surgical resection
* Tumor lesion is 5-15 cm from anal verge
* cT2 N+ or cT3-T4 N0 or N+ as assessed by endorectal ultrasound scan (US)
* No evidence of distant metastatic disease
* Signed informed consent prior to initiation of any study-specific procedure or treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Able to comply with the protocol, including tissue sampling, imaging studies and surgical intervention
* Life expectancy more than 12 weeks
* Absolute neutrophil count >= 1500 per mm^3
* Platelet count >= 100,000 per mm^3
* Hemoglobin >= 9 g/dL (may be transfused to maintain or exceed this level)
* Total bilirubin < 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase and alanine aminotransferase < 2.5 x ULN
* Calculated creatinine clearance according to Cockroft and Gault formula >= 50 mL/min
* Urine for proteinuria should be < 2 +; patients discovered to have >= 2 + proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 1 g of protein in 24 hours
* International normalized ratio =< 1.5 and activated prothrombin time =< 1.5 x ULN within 7 days prior to enrollment; the use of full-dose oral or parenteral anticoagulants is permitted as long as the international normalized ratio (INR) or activated partial thromboplastin time (aPTT) is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least two weeks prior to the first study treatment
* Female patients should not be pregnant or breast-feeding. Female patients, if not postmenopausal (< 12 months of amenorrhea) or surgically sterile, should agree to use effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) during the study and for a period of at least 6 months following the last administration of study drugs. Female patients with an intact uterus (unless amenorrheic for the last 24 months) must have a negative serum pregnancy test within 7 days prior to randomization into the study
* Fertile male patients must agree to use a highly effective contraceptive method (i.e., with a failure rate of < 1 % per year, such as vasectomy, sexual abstinence, or female partner's use of hormonal implants or combined oral contraceptives) during the trial and for a period of at least 6 months after the last dose of study drug
* Archival tumor tissue sample must be requested and available prior to study entry; a copy of the local pathology report must be submitted along with the specimens; patients without available archival tissue are excluded

Exclusion Criteria:

* Prior chemotherapy or radiotherapy for colorectal cancer
* Clinical evidence of bleeding diathesis or coagulopathy
* Pregnancy or lactation
* Sensory peripheral neuropathy >= grade 2
* Known positivity for human immunodeficiency virus (HIV)
* Malignancies other than rectal cancer within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, and ductal carcinoma in situ treated surgically with curative intent
* Radiotherapy to any site for any reason within 28 days prior to study entry
* Treatment with any other investigational agent, or participation in another investigational drug trial within 28 days prior to randomization
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding, or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of bevacizumab or puts the patient at high risk for treatment-related complications
* Surgery (including open biopsy), significant traumatic injury within 28 days prior to randomization, minor surgery, including insertion of an indwelling catheter, within 24 hours prior to the first bevacizumab infusion is allowed
* Current or recent (within 10 days prior to first dose of bevacizumab) use of aspirin (> 325 mg/day)
* History or evidence of inherited bleeding diathesis or coagulopathy with a risk of bleeding
* Inadequately controlled hypertension (blood pressure: systolic > 150 mmHg and/or diastolic > 100 mmHg)
* Clinically significant (i.e., active) cardiovascular disease (e.g., cerebrovascular accident or myocardial infarction within 6 months prior to randomization), unstable angina, congestive heart failure (New York Heart Association Class >= II) or serious cardiac arrhythmia that is uncontrolled by medication or may interfere with administration of study treatment
* Serious non-healing wound, active peptic ulcer, or untreated bone fracture
* History of abdominal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months of randomization
* Known hypersensitivity to bevacizumab or any of its excipients or any other study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-08-02 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2023-06-24 (Estimated)

PRIMARY OUTCOMES:
Rate of CPR in the pathology specimen | Up to 3 years

SECONDARY OUTCOMES:
Tumor regression on mesorectal margins (pathologic stage lower than clinical stage) | Up to 3 years
Rate of locoregional recurrence | Up to 3 years
Incidence and nature of adverse events (AEs) according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 ( v4) | Up to 3 years
Incidence and nature of serious AEs (SAEs) according to NCI CTCAE v4.0 | Up to 3 years
Incidence and nature of AEs of special interest for bevacizumab (grades) according to NCI CTCAE v4.0 | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Afsaneh Barzi, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Barzi A, Choi A, Tsao-Wei D, Iqbal S, El-Khoueiry A, Agafitei DR, Cologne KG, Lenz HJ. Phase II Trial of Neoadjuvant Bevacizumab with Modified FOLFOX7 in Patients with Stage II and III Rectal Cancer. Oncologist. 2020 Dec;25(12):e1879-e1885. doi: 10.1634/theoncologist.2020-0642. Epub 2020 Aug 27. PMID 32649004